CLINICAL TRIAL: NCT02665624
Title: Adding Stewed Apricot Juice to Senna Improves the Right-Side and Overall Colon Cleansing Quality for Colonoscopy Preparation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Camlıca Erdem Hospital (Other)
Responsible Party: Principal Investigator, Bulent Yasar, M.D., Camlıca Erdem Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: HNEAH-2015/KK/04
Record Dates: First submitted 2016-01-16; First posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Colonoscopy Preparation
Keywords: Bowel cleansing; Colonoscopy; Stewed apricot juice; Senna
MeSH Terms: interventions — Sennosides

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stewed apricot juice + senna group (Active Comparator): 68 patients received 250 ml of Senna solution (containing 500 mg sennoside A+B calcium) (X-M solution, Yenisehir Pharmaceuticals, Turkey) at 6 PM on the day before colonoscopy, and at 6 AM on the day of the procedure. Additional one liter of stewed apricot juice (made with dried apricot) were told to be drunken until 2 h before colonoscopy.
  Interventions: Drug: Senna and stewed apricot juice
- senna alone group (Active Comparator): 60 patients received 250 ml of Senna solution (containing 500 mg sennoside A+B calcium) (X-M solution, Yenisehir Pharmaceuticals, Turkey) at 6 PM on the day before colonoscopy, and at 6 AM on the day of the procedure. 1 patient was dropped out due to obstructive sigmoid colon cancer.
  Interventions: Drug: Senna alone

INTERVENTIONS:
Drug: Senna and stewed apricot juice — comparison of bowel cleansing and patient comfort.
  Other Names: X-M solution (300 mg sennoside A+B calcium, Yenisehir Pharmaceuticals); Stewed apricot juice made with dried apricot
  Arms: Stewed apricot juice + senna group
Drug: Senna alone — comparison of bowel cleansing and patient comfort.
  Other Names: X-M solution (300 mg sennoside A+B calcium, Yenisehir Pharmaceuticals)
  Arms: senna alone group

SUMMARY:
Adequate bowel cleansing is essential for optimal colonoscopic examination. However, none of the colonoscopy preparation regimens is safe, efficient and also comfortable. The investigators' aim was to determine whether adding stewed apricot juice to senna increases patient comfort and improves bowel cleansing during colonoscopy preparation.

DETAILED DESCRIPTION:
* Colonoscopy is the current standard method for diagnosing colon cancer and polyps, and also can be used for therapeutic interventions such as polypectomy. Diagnostic accuracy and therapeutic safety of the procedure depends on the quality of the colonic cleansing. Inadequate bowel preparation may result in missed precancerous lesions, longer colonoscopy time, lower cecal intubation rates and increased electrocautery risks. It also causes further costs because the colonoscopy has to be re-scheduled or alternative examinations have to be planned.
* Although polyethylene glycol (PEG) and sodium phosphate (NaP) are the main cleansing solutions in current practice, they tend to be poorly tolerated. The need to intake a large volume of fluid and unpleasant, salty taste of PEG reduce patient compliance. To overcome these limitations, split-dose administration of PEG has been shown effective and more patient-friendly. Unfortunately, PEG solutions have not been available in some countries due to marketing problems, as in Turkey. The potential risks for clinically significant alterations in serum electrolyte levels and hemodynamic instability in patients with renal failure, congestive heart failure, uncontrolled hypertension and ascites limits the usage of NaP. Moreover, European Society of Gastrointestinal Endoscopy (ESGE) suggests that oral NaP can only be advised in selected cases such as patients unable to tolerate other agents or only individuals to be at low risk of NaP-related side-effects. Unfortunately, 20% of patients who consumed PEG or NaP did not have satisfactory bowel cleansing. Because of the limitations of NaP and unavailability of PEG solutions, senna is still the main colonoscopy preparation in some countries..
* The ideal colonoscopy preparation would not only reliably empty the colon, but also not cause any patient discomfort. However, none of the preparations currently meet all of these criteria. Thus, numerous clinical trials have assessed prokinetic and spasmolytic agents, ascorbic acid, olive oil, orange and pineapple juice to attempt to improve the effectiveness and tolerance of colonoscopic preparation regimens. Among these preparations, no additive effect was demonstrated for prokinetic and spasmolytic agents, while authors determined more patient satisfaction and colon cleansing for the rest.
* Senna alkaloids have a direct effect on intestinal mucosa, increasing the colonic motility, enhancing colonic transit, and inhibiting water and electrolyte secretion. Although senna were used effectively alone in the past, they have been replaced by PEG and NaP solutions. Senna have a good-taste and are well-tolerated, inexpensive and have fewer adverse effects, yet, their efficacy is controversial.
* Apricot (Prunus armeniaca L.) has an important place in human nutrition and can be used as fresh or dried. Also, traditionally dried apricots have been used for many years in Mediterranean countries as a remedy for constipation because of their high-fiber content . Furthermore, apricots contain sorbitol (4,6g/100g) which has a laxative effect and used for treating constipation in the elderly.
* Although these fruits are already in our life, to investigators knowledge, there is no study examining the effects of apricot juice for precolonoscopic preparation. Therefore, the investigators conducted this study to establish whether adding stewed apricot juice to senna promotes bowel cleansing as well as patient comfort.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with either sex who were over 18 years of age and referred for elective colonoscopy were included in the study

Exclusion Criteria:

* history of renal, cardiac, hepatic and metabolic disease including diabetes mellitus
* history of colonic resection
* hospitalized patients
* pregnancy or breast-feeding
* history of inflammatory bowel disease
* known allergy to senna.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The quality of overall colon cleansing | During colonoscopy
  The quality of colon cleansing was evaluated by using the validated Ottawa Bowel Preparation Quality Scale (Table 1). The score was calculated by adding the 0 to 4 ratings for recto-sigmoid, transverse and right colon separately and the 0 to 2 fluid quantity rating. 0, 1 and 2 scores were accepted for adequate preparation while 3 and 4 not, for each colonic segment.
  Table 1 Ottawa Bowel Preparation Quality Scale Score Description 0 No fluid
  1. Able to see mucosa without aspiration
  2. Able to see mucosa after aspiration
  3. Able to see mucosa after both washing and aspiration
  4. Solid stool, incapable of aspiration

SECONDARY OUTCOMES:
The quality of cleansing in the right colon, and patient comfort. | During colonoscopy and the day before colonoscopy, respectively.
  0, 1 and 2 scores were accepted for adequate preparation while 3 and 4 not, for right colonic segment.
  Upon arrival at the endoscopy unit,the participants were asked to complete a nurse-administered questionnaire to assess their tolerability and adverse events during preparation. This questionnaire included of 18 questions and was used in similar previous studies specified in references section.
  Participant acceptability was assessed as difficulty of finishing ingestion of the regimens.
  Participant compliance was defined as success in consuming the total amount of the regimens.
  Participants were also asked for willingness to receive the same regimen in the future.
  Participants were assessed for safety based on frequency and severity of adverse events nausea, vomiting, abdominal pain, abdominal bloating, weakness,sleep disturbance and anal irritation symptoms rated for absent, mild, moderate and severe.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Aronchick CA, Lipshutz WH, Wright SH, Dufrayne F, Bergman G. A novel tableted purgative for colonoscopic preparation: efficacy and safety comparisons with Colyte and Fleet Phospho-Soda. Gastrointest Endosc. 2000 Sep;52(3):346-52. doi: 10.1067/mge.2000.108480. PMID 10968848
- [Result] Abut E, Guveli H, Yasar B, Bolukbas C, Bolukbas FF, Ince AT, Kendir T, Dalay AR, Kurdas OO. Administration of olive oil followed by a low volume of polyethylene glycol-electrolyte lavage solution improves patient satisfaction with right-side colonic cleansing over administration of the conventional volume of polyethylene glycol-electrolyte lavage solution for colonoscopy preparation. Gastrointest Endosc. 2009 Sep;70(3):515-21. doi: 10.1016/j.gie.2009.01.002. Epub 2009 Jun 24. PMID 19555936
- [Result] Berkelhammer C, Ekambaram A, Silva RG. Low-volume oral colonoscopy bowel preparation: sodium phosphate and magnesium citrate. Gastrointest Endosc. 2002 Jul;56(1):89-94. doi: 10.1067/mge.2002.125361. PMID 12085041